CLINICAL TRIAL: NCT01139385
Title: Comparative Study Between Clipless Laparoscopic Cholecystectomy Using Harmonic Scalpel Versus Conventional Method in Day Surgery: a Prospective Randomized Study
Brief Title: Clipless Laparoscopic Cholecystectomy Using Harmonic Scalpel Versus Conventional Method in Day Surgery
Acronym: CLCHS
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Saverio Mari, Reserch Fellows, University of Roma La Sapienza
Other Study IDs: DS-001
Record Dates: First submitted 2010-06-02; First posted 2010-06-08 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2013-12

CONDITIONS: Cholelithiasis
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- clipless: laparoscopic cholecystectomy performed by harmonic scalpel with closure and division of the cystic duct only by the device
  Interventions: Procedure: Harmonic scalpel
- traditional: laparoscopic cholecystectomy performed by harmonic scalpel with closure of the cystic duct only by titanium clip
  Interventions: Procedure: Traditional

INTERVENTIONS:
Procedure: Harmonic scalpel — The Cholecystectomy is performed using only Harmonic Scalpel to mobilize the Cholecystis and to close the cystic duct and the cystic artery
  Groups: clipless
Procedure: Traditional — The cholecystectomy is performed using Harmonic Scalpel to mobilize the cholecystis and the cystic duct and the cystic artery are closed by titanium clips
  Groups: traditional

SUMMARY:
The aim of this study was to compare between the safety and efficacy of the harmonic shears and the commonly used clip technique in achieving safe closure and division of the cystic duct in the laparoscopic cholecystectomy in day surgery setting

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Cholelithiasis
* Age under 65 yr old
* BMI under 35
* ASA I or II

Exclusion Criteria:

* Acute cholecystitis
* Suspect of common bile duct stones

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with gallstone undergoing cholecystectomy in day surgery setting
Sampling Method: Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2008-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
effectiveness closure of the cystic duct | at 1 months
  the effectiveness closure of the cystic duct is assessed on the presence or not of cystic duct bile leak

SECONDARY OUTCOMES:
postoperative complication | 1 month
  the presence of postoperative complication is investigated
efficacy and safety of the use of harmonic scalpel performing cholecystectomy | 24 hours
  the efficacy and safety of the use of harmonic scalpel performing cholecystectomy is assessed by evaluating the operative time, the presence of major or minor intraoperative complication and the postoperative complication.

CONTACTS AND LOCATIONS:
Locations (1):
- Oneday - Day Surgery Unit - Azienda Ospedaliera Sant'Andrea - University Sapienza of Rome, Rome, Italy, Italy